CLINICAL TRIAL: NCT00147615
Title: Peds II (Pediatric Eplerenone Development Study II)--An Open Label, Long-Term Study To Evaluate The Safety Of Eplerenone In The Treatment Of Hypertension In Children
Brief Title: The Long-term Study to Evaluate the Safety of Eplerenone in the Treatment of Hypertension in Children Aged 6 to 16 Years
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A6141077
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Eplerenone

INTERVENTIONS:
Drug: Eplerenone

SUMMARY:
To assess the long-term safety and toleration of eplerenone in the children aged 6 to 16 years with high blood pressure. The study will last at least 1 year and about 140 patients will participate.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 6 to 16 years
* The seated systolic blood pressure greater than or equal to the 95th percentile for age, gender and height, measured on at least 3 separate occasions

Exclusion Criteria:

* K/DOQI classification of stages of chronic kidney disease equal to 4 or 5
* Serum or whole blood potassium > 5.5. mEq/L

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140
Dates: Start 2004-10; Study Completion 2006-06

PRIMARY OUTCOMES:
Safety of eplerenone in hypertensive children

SECONDARY OUTCOMES:
Efficacy and pharmacokinetics of eplerenone in hypertensive children

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (15):
- United States (6):
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Park Ridge, Illinois
  - Pfizer Investigational Site, Durham, North Carolina
  - Pfizer Investigational Site, Columbus, Ohio
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Katy, Texas
- India (6):
  - Pfizer Investigational Site, Hyderabad, Andhra Pradesh
  - Pfizer Investigational Site, Bangalore, Karnataka
  - Pfizer Investigational Site, Chennai, Tamil Nadu
  - Pfizer Investigational Site, Chennai
  - Pfizer Investigational Site, Mumbai
  - Pfizer Investigational Site, New Delhi
- Russia (3):
  - Pfizer Investigational Site, Moscow
  - Pfizer Investigational Site, Saint Petersburg
  - Pfizer Investigational Site, Smolensk

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6141077&StudyName=The+long%2Dterm+study+to+evaluate+the+safety+of+Eplerenone+in+the+treatment+of+hypertension+in+children+aged+6+to+16+years